CLINICAL TRIAL: NCT06491615
Title: National Ophthalmic Genotyping and Phenotyping Network, Stage 3 - Expansion of DNA and Data Repositories for Rare Inherited Ophthalmic Diseases
Brief Title: National Ophthalmic Genotyping and Phenotyping Network (eyeGENE (Registered Trademark)), Stage 3 - Expansion of DNA and Data Repositories for Rare Inherited Ophthalmic Diseases
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001647; 001647-EI
Record Dates: First submitted 2024-07-08; First posted 2024-07-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08-15

CONDITIONS: Inherited Ophthalmic Diseases; Hypopigmentation Disorder; Corneal Dystrophy; Blue-cone Monochromacy; Best Disease; Aniridia; Albinism
Keywords: eyeGENE; Genetics; Inherited
MeSH Terms: conditions — Vitiligo; Corneal Dystrophies, Hereditary; Blue cone monochromatism; Vitelliform Macular Dystrophy; Aniridia; Albinism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants with inherited eye diseases or relative of affected participant

SUMMARY:
Background:

The eyeGENE (Registered Trademark) program is a research resource for inherited eye conditions which includes genotypic and phenotypic data, imaging, and a corresponding biobank of DNA samples from people with a variety of eye diseases. Since 2007 this registry has been helping researchers learn more about the genetic sources for many inherited eye diseases. These findings helped them create better treatments. Now researchers want to expand eyeGENE (Registered Trademark) to include more people for certain eye diseases.

Objective: To collect information and DNA samples for the study of eye diseases.

* Primary objective

  --To expand the current eyeGENE (Registered Trademark) data repository with targeted participant accrual
* Secondary objectives

  * To enhance recruitment for clinical trials and investigations in inherited eye diseases

    * To establish genotype-phenotype correlations for rare eye diseases

Eligibility:

People of any age with certain eye diseases. These can include aniridia; Best disease; blue-cone monochromacy; corneal dystrophy; and disorders of pigmentation, such as albinism. Relatives unaffected by the eye disease of interest may also be needed.

Design:

Researchers will select participants based on their diagnosis. The data may include images and test results from eye exams.

Participants will provide a sample of saliva. They will receive a kit with written instructions. They will spit in a tube and mail it to the NIH.

Participants may be asked to provide a blood sample. The blood may be drawn at the NIH or at a local clinic.

The eyeGENE (Registered Trademark) repository will offer researchers data about the participants eye conditions. The data may include pictures of their eyes, results of the genetic testing, and history of other diseases. Researchers will be able to see data such as age and gender, but they will not see names, dates of birth, or contact information.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

Molecular genetics has revolutionized the diagnosis and treatment of inherited eye diseases. Progress in research on inherited eye disease is augmented by the availability of patient DNA coupled to phenotypic information. To expand the current eyeGENE (Registered Trademark) data repository, participants will be accrued from targeted rare and ultra-rare disease populations.

OBJECTIVES:

Primary Objective:

-To expand the current eyeGENE (Registered Trademark) data repository with targeted participant accrual

Secondary Objectives:

* To enhance recruitment for clinical trials and investigations in inherited eye diseases
* To establish genotype-phenotype correlations for rare eye diseases

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

The participant must present with characteristics consistent with one of the following diagnoses:

* Aniridia
* Best disease
* Blue-cone monochromacy
* Corneal dystrophy
* Other hypopigmentation disorder affecting vision (e.g., Oculocutaneous and ocular albinism, Hermansky-Pudlak syndrome, Chediak-Higashi syndrome)

OR

The participant must be a direct, close relative of an affected participant.

OR

A participant who also participated in the eyeGENE Stage 1 protocol who may benefit from further genetic testing.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Those with impaired decision-making capability who do not have a legally-authorized representative.
* Those unable to provide a saliva sample OR have any disease or condition that makes it unsafe for a subject to provide a suitable blood sample of at least 5 mL to yield more than 50 micrograms of DNA.

An individual who meets any of the following criteria will be excluded from participation in the optional retinal imaging:

* Those with a history of epilepsy.
* Children under the age of 18.

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with inherited eye diseases or their unaffected relatives.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2054-06-27 (Estimated); Study Completion 2054-06-27 (Estimated)

PRIMARY OUTCOMES:
To expand the current eyeGENE data repository with targeted participant accrual. | 30 years
  To expand the current eyeGENE data repository with targeted participant accrual.

SECONDARY OUTCOMES:
To enhance recruitment for clinical trials and investigations in inherited eye diseases. | 30 years
  To enhance recruitment for clinical trials and investigations in inherited eye diseases.
To establish genotype-phenotype correlations for rare eye diseases. | 30 years
  To establish genotype-phenotype correlations for rare eye diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- United States (2):
  - National Eye Institute (NEI), Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001647-EI.html